CLINICAL TRIAL: NCT05027191
Title: Evaluating the Effect of Desflurane Versus Sevoflurane With Recent Biomarkers of Renal and Hepatic Function in Laparoscopic Cholecystectomy Patients: A Prospective Randomized Double Blinded Study
Brief Title: Effect of Desflurane Versus Sevoflurane With Recent Bio-markers on Renal and Hepatic Functions
Status: Completed | Type: Observational
Sponsor: Theodor Bilharz Research Institute (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, khalda Galal Moustafa, Principal Investigator, Theodor Bilharz Research Institute
Other Study IDs: 110-T
Record Dates: First submitted 2019-09-11; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Sevoflurane: This group will receive sevoflurane as the maintenance inhalational anesthetic.
  Interventions: Diagnostic Test: Neutrophil Gelatinase-Associated Lipocalin (NGAL); Drug: Sevoflurane
- Desflurane: This group will receive desflurane as the maintenance inhalational anesthetic.
  Interventions: Diagnostic Test: Neutrophil Gelatinase-Associated Lipocalin (NGAL); Drug: Desflurane

INTERVENTIONS:
Diagnostic Test: Neutrophil Gelatinase-Associated Lipocalin (NGAL) — The evaluation of inhalational anesthetics (desflurane and sevoflurane) on NGAL levels in laparoscopic cholecystectomy patients.
Drug: Desflurane — Desflurane
  Groups: Desflurane
Drug: Sevoflurane — Sevoflurane
  Groups: Sevoflurane

SUMMARY:
Studying the effects of both inhalational anesthetics desflurane and sevoflurane on hepatic integrity and renal function, guided by recent blood and urine biomarkers in patients undergoing laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Class: I&II.
2. Elective laparoscopic cholecystectomy.
3. Age: 25-55 years.
4. Gender: Both male and female.
5. Body Mass Index (BMI): 18.5-24.9 km2-(Normal weight).

Exclusion Criteria:

1. Extremes of age.
2. Abnormal hepatic function by alanine aminotransferase (ALT) and aspartate aminotransferase (AST) values outside the normal range.
3. Abnormal renal function by blood urea nitrogen (BUN) and creatinine above the normal ranges.
4. Hypertension, unstable angina pectoris or myocardial infarction within the last six months.
5. Pregnancy and lactation.
6. Bronchial asthma.
7. Drug allergies.
8. Alcohol or drug addiction.
9. General anesthesia within the last three months.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: After informed written consents have been taken, this study will be conducted on 70 patients scheduled for laparoscopic cholecystectomy. The patients will be randomly allocated into two groups (a desflurane (D) group and a sevoflurane (S) group) using a sealed envelope technique for each group.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in serum Neutrophil gelatinase-associated lipocalin (NGAL) | a change from baseline NGAL serum level at 6 hours
  Renal Biomarker

SECONDARY OUTCOMES:
Change in serum Arginase | Baseline, first hour, six hours, after 24 hours
  Hepatic biomarker
Change in serum Cystatin-c | Baseline, first hour, six hours, after 24 hours
  Hepatic biomarker
Change in urine Netrin-1 | Baseline, first hour, six hours, after 24 hours
  Renal biomarker
Change in urine Kidney Injury Molecule | Baseline, first hour, six hours, after 24 hours
  Renal biomarker
Change in urine Interleukin-18 | Baseline, first hour, six hours, after 24 hours
  cytokines
Change in urine Alpha-Glutathione S-Transferase | Baseline, first hour, six hours, after 24 hours
  Liver biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Khalda G Radwan, MD, Principal Investigator — Theodor Bilharz Rsearch Institute
Locations (1):
- Theodor Bilharz Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided